CLINICAL TRIAL: NCT02535377
Title: Molecular Diagnostic of Sperm Cryoresistance of Semen Donors and Clinical Outcomes After Artificial Insemination. Optimization of Sperm Bank
Brief Title: Human Sperm Markers of Cryodamage Resistance
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Collaborators: Igenomix (Industry)
Responsible Party: Principal Investigator, Elena Sellés Soriano, Molecular diagnostic of sperm cryoresistance of semen donors and clinical outcomes after artificial insemination. Optimization of sperm bank, Instituto Valenciano de Infertilidad, IVI Alicante
Other Study IDs: 1406-ALC-048-ES
Record Dates: First submitted 2015-07-02; First posted 2015-08-28 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2020-01

CONDITIONS: Fertility
Keywords: Cryodamage; microarrays; Insemination; sperm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High cryoresistance: High resistance to sperm cryopreservation (decreased sperm motility <20%)
  Interventions: Other: Sperm cryopreservation
- Low cryoresistance: Low resistance to sperm cryopreservation (decreased sperm motility >20%)
  Interventions: Other: Sperm cryopreservation

INTERVENTIONS:
Other: Sperm cryopreservation — Sperm from the different groups are cryopreserved to evaluate their resistance to preservation.

SUMMARY:
Sperm freezing has been employed for decades for male fertility preservation in cases of foreseeable or unexpected loss of fertility to guarantee future paternity, and also as a complement of assisted reproduction techniques.

Sperm quality after thawing is highly variable, even among consecutive samples from the same individual, with mean survival rates around 40%. To date, the molecular basis of the adequate resistance or intolerance to freezing/thawing protocols is unknown, and its knowledge can lead to improvement in the selection of the samples to be frozen and also in the adequate supplement of cryopreservation media. Microarray analysis provides a powerful tool to address the molecular explanation beyond this behaviour, yielding results about comparative messenger ribonucleic acid (mRNA)expression under the two different biological conditions: optimal and suboptimal survival.

Then, the aim of the investigators' study is to determine the genomic profile of sperm samples depending on their survival resistance to cryopreservation, to determine genes involved in cryodamage sensitivity.

DETAILED DESCRIPTION:
Nested cases and controls design, with donor sperm samples frozen under conventional protocols, categorized depending on their good (GSR, n=20) (less than 20% motility decrease) or bad (BSR, n=20) (more than 20% motility decrease) survival rates. Sperm mRNA was extracted using Trizol protocol, suspended in diethylpyrocarbonate (DEPC)-treated water and frozen at -80 degrees until the microarray experiments were performed. RNAs were analyzed on Agilent Bioanalyzer 2100. Samples were pooled in 4 (5 samples/pool and 4 pools/group). Finally, 8 Agilent One colour Whole genome microarray (44K) were performed with pooled samples, 4 microarrays per group.

The results will be evaluate to detect those genes differentially expressed.

ELIGIBILITY:
Inclusion Criteria:

The criteria used for the inclusion of donors in the sperm bank will be considered:

* males from 18 to 35 years.
* good physical and psychological conditions and no hereditary diseases
* seminal parameters: concentration > 40 million sperm / ml; percentage of progressive motility> 50% percentage of normal forms> 4%.
* For pregnancy rates after artificial insemination, only women< 40 years without tubal pathologies and artificial insemination indications will be included.

Exclusion Criteria:

All the population not included in the list of inclusion will be excluded.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men from 18-35 years, included in the donation program of IVI Alicante. Any transmisible clinical pathology, viral infection or genetic disease should be ruled out by family history records.
  In addition, seminal samples from donors must meet the seminal criteria considered by our laboratory:
  * sperm concentration> 40 million sperm / ml;
  * percentage of progressive motility> 50%
  * percentage of normal forms> 4%.
  For pregnancy rates after IUI, only women< 40 years without tubal pathologies and IUI indications will be included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02-12; Primary Completion 2018-11-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Genomic profile of sperm samples depending on their survival resistance to cryopreservation | A year and a half
  The genomic profile of sperm samples depending on their survival resistance to cryopreservation will be analysed and expressed as:
  * Common or differentially expressed genes: in case of genes expressed in both groups
  * Exclusive Genes, in case of genes expressed just in one group

SECONDARY OUTCOMES:
Pregnancy rates after artificial insemination with donor semen in the different groups. | two years
  Once obtained the genomic profile of samples from donors included the different groups, we will analyze its relationship with the reproductive outcomes, in particular pregnancy rates after conventional artificial insemination (percentage of positive pregnancy test)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sellés, PhD, Principal Investigator — Instituto Valenciano de Infertilidad, IVI Alicante
Locations (1):
- IVI Alicante, Alicante, Spain

REFERENCES:
- [Background] Thurston LM, Siggins K, Mileham AJ, Watson PF, Holt WV. Identification of amplified restriction fragment length polymorphism markers linked to genes controlling boar sperm viability following cryopreservation. Biol Reprod. 2002 Mar;66(3):545-54. doi: 10.1095/biolreprod66.3.545. PMID 11870056
- [Background] Thurston LM, Watson PF, Holt WV. Semen cryopreservation: a genetic explanation for species and individual variation? Cryo Letters. 2002 Jul-Aug;23(4):255-62. PMID 12391486
- [Background] Holt WV, Medrano A, Thurston LM, Watson PF. The significance of cooling rates and animal variability for boar sperm cryopreservation: insights from the cryomicroscope. Theriogenology. 2005 Jan 15;63(2):370-82. doi: 10.1016/j.theriogenology.2004.09.018. PMID 15626405
- [Background] Casas I, Sancho S, Briz M, Pinart E, Bussalleu E, Yeste M, Bonet S. Freezability prediction of boar ejaculates assessed by functional sperm parameters and sperm proteins. Theriogenology. 2009 Oct 15;72(7):930-48. doi: 10.1016/j.theriogenology.2009.07.001. Epub 2009 Aug 3. PMID 19651432
- [Background] Garrido N, Martinez-Conejero JA, Jauregui J, Horcajadas JA, Simon C, Remohi J, Meseguer M. Microarray analysis in sperm from fertile and infertile men without basic sperm analysis abnormalities reveals a significantly different transcriptome. Fertil Steril. 2009 Apr;91(4 Suppl):1307-10. doi: 10.1016/j.fertnstert.2008.01.078. Epub 2008 Mar 25. PMID 18367176
- [Background] Garcia-Herrero S, Meseguer M, Martinez-Conejero JA, Remohi J, Pellicer A, Garrido N. The transcriptome of spermatozoa used in homologous intrauterine insemination varies considerably between samples that achieve pregnancy and those that do not. Fertil Steril. 2010 Sep;94(4):1360-1373. doi: 10.1016/j.fertnstert.2009.07.1671. Epub 2009 Sep 30. PMID 19796764
- [Background] Garcia-Herrero S, Garrido N, Martinez-Conejero JA, Remohi J, Pellicer A, Meseguer M. Ontological evaluation of transcriptional differences between sperm of infertile males and fertile donors using microarray analysis. J Assist Reprod Genet. 2010 Feb;27(2-3):111-20. doi: 10.1007/s10815-010-9388-5. Epub 2010 Feb 2. PMID 20127162
- [Background] Rahana AR, Ng SP, Leong CF, Rahimah MD. Comparison between mechanical freezer and conventional freezing using liquid nitrogen in normozoospermia. Singapore Med J. 2011 Oct;52(10):734-7. PMID 22009393
- [Background] Gadea J, Molla M, Selles E, Marco MA, Garcia-Vazquez FA, Gardon JC. Reduced glutathione content in human sperm is decreased after cryopreservation: Effect of the addition of reduced glutathione to the freezing and thawing extenders. Cryobiology. 2011 Feb;62(1):40-6. doi: 10.1016/j.cryobiol.2010.12.001. Epub 2010 Dec 13. PMID 21156167